CLINICAL TRIAL: NCT00991406
Title: Neural Prostheses and Gait Performance: Model-Based Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4668-R
Record Dates: First submitted 2009-10-02; First posted 2009-10-08 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-07

CONDITIONS: Hemiplegia
Keywords: Electric Stimulation; Hemiplegia; walking
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: FES (Experimental): Case-control study: pre- and post-stimulation (FES).
  Interventions: Device: FES

INTERVENTIONS:
Device: FES — Surface stimulation to contract the muscles in the lower extremity

SUMMARY:
The purpose of this research is to find the optimal patterns of functional electrical stimulation (FES) of muscles in the lower legs that will improve walking ability in those who have had a stroke and at the same time ensure walking stability. FES involves applying small electric currents to the nerves, which cause the muscles to contract.

FES research projects vary from simple investigations of the therapeutic effects of exercise on muscle function and skin health, to more complex studies of functional movements such as standing or walking.

DETAILED DESCRIPTION:
The study aims to find the optimal patterns of functional electrical stimulation (FES) of muscles in the lower legs that will improve walking ability in those who have had a stroke and at the same time ensure walking stability will be achieved through an analytical approach comprised of computational models and gait simulations to objectively determine patient-specific patterns of muscle activation. The investigators will develop a computer simulation of the dynamics of hemiplegic gait characterized by unilateral plantarflexor weakness. Then, the investigators will relate the results of the computer model results to real data collected from subjects with known plantarflexor weakness to provide a theoretical basis for improving gait efficiency and stability with FES.

ELIGIBILITY:
Inclusion Criteria:

This study includes stroke survivors greater than 18 years of age, >180 days from first clinical hemorrhagic or nonhemorrhagic stroke with:

* Unilateral hemiparesis with sufficient endurance and motor ability to ambulate >30 feet continuously without an AFO requiring no more than 25% physical help
* Berg Balance Scale score >23 without assistive devices
* Standing ankle dorsiflexion strength of <4/5
* Foot-drop during ambulation with gait instability or inefficient gait defined as supervision need
* Possible use of physical assistance or assistive device (cane, walker)
* Evidence of foot-drop as seen by "dragging" or "catching" of affected toes during limb swing or circumducting affected limb
* Vaulting of the unaffected limb or hiking the affected hip to clear toes.
* Intact and electrically ex-citable lower motor neurons
* Ankle dorsiflexion to at least neutral while standing with electrical stimulation of common peroneal and tibial nerves without painful hypersensitivity to stimulation
* Adequate social support and stability
* Medically stable with intact skin in affected lower limb
* Willingness to comply during research procedures
* No systemic co-morbidities
* No history of potentially fatal cardiac arrhythmias i.e. ventricular tachycardia, supraventricular tachycardia and rapid ventricular response atrial fibrillation with hemodynamic instability
* No psychological problems or chemical dependency
* No acute medical complications such as depression or chronic anxiety requiring long term pharmacological therapy. Able-bodied controls must be of similar age, body mass and stature as those with hemiparesis and must be free of any medical and disabling orthopedic problems.

Exclusion Criteria:

In addition to failure to meet the inclusion criteria, participants will be excluded from the study for the following:

* Requires an ankle foot orthosis (AFO) to prevent knee flexion collapse in stance
* Excessive edema of affected extremity
* Absent sensation in affected limb
* History of potentially fatal cardiac arrhythmias such as ventricular tachycardia, supraventricular tachycardia, and rapid ventricular response, atrial fibrillation with hemodynamic instability
* Demand pacemakers or any implanted electronic systems
* Pregnancy
* Uncontrolled seizure disorder
* Ipsilateral lower limb lower motor neuron lesion
* Parkinson's disease
* Spinal cord injury
* Traumatic brain injury
* Multiple sclerosis
* Ankle plantar flexor contraction
* Severely impaired cognition and communication
* Painful hypersensitivity to neuromuscular stimulation of common peroneal nerve
* Knee hyperextension (genu recurvatum) that cannot be adequately corrected with peroneal nerve stimulation
* History of botulinum toxin to the lower extremity within the prior three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Hardin van den Bogert, PhD MS, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Computational optimization was via tracking joint angles & ground reaction forces from an able walking subject.We optimized the hemiparetic (HP) subject's model to able data & their walking data producing optimization solutions for muscle activations in each case.The able subject was not considered enrolled,only 9 HPsubjects were actually enrolled.
Period: Overall Study
Arm/Group | Arm 1: FES
Started | 9
Completed | 8 (One participant did not respond to FES due to tone.)
Not Completed | 1
Not completed — One participant did not respond to FES. | 1

BASELINE CHARACTERISTICS:
Population: The able-bodied participant was only used to develop the computational optimization and was not considered to be enrolled in the study.
Groups:
- Arm 1: FES: Case-control study: pre- and post-stimulation (FES).
  FES: Surface stimulation to contract the muscles in the lower extremity where subjects serve as their own control.
Arm/Group | Arm 1: FES
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Walking Stability and Speed
Description: This was a feasibility study of computational models and gait simulations to objectively determine patient-specific patterns of muscle activation. We developed computer models and walking simulations of hemiplegic gait from 8 subjects. We related the model results (muscle activations) to the optimized data collected from hemiplegic subjects & calculated the FES pattern to be delivered in 2 forms (open loop & foot switch triggered). The primary outcome measure turned out to be the feasibility of the methods because after developing our computer modeling and computational optimization framework we could only test walking with the 2 forms of FES at the same preferred walking speed on a treadmill. Thus, the simulated walking speed and the real walking speed pre and post FES turned out to be the same. Walking stability was measured with variability in work performed at the ankle. The additional volitional and FES biomechanical data that were measured are listed in the secondary measures.
Time Frame: pre-stimulation (volitional) and post-stimulation (FES), day of the study
Population: Volitional and FES data available for participants with hemiparesis.
Measure: Mean (Standard Deviation); unit: Joules/body mass in kilograms
Arm/Group | Arm 1: FES
Number analyzed (Participants) | 8
Joules/body mass in kilograms
  Volitional | 0.1055 (0.0117)
  FES: Open loop | 0.0390 (0.0716)
  FES: Foot switch Trigger | 0.0206 (0.0209)

2. Secondary Outcome: Peak Ankle Power
Description: This is the peak ankle power during walking normalized by body weight.
Time Frame: Same day: pre-stimulation (volitional) and post-stimulation (FES), day of the study
Population: Volitional and FES data available for participants with hemiparesis.
Measure: Mean (Standard Deviation); unit: Watts/body mass in kilograms
Arm/Group | Arm 1: FES
Number analyzed (Participants) | 8
Watts/body mass in kilograms
  Volitional | 0.9162 (1.0242)
  FES: Open Loop | 1.1392 (1.1438)
  FES: Foot switch Trigger | 0.6315 (0.6106)

3. Secondary Outcome: Positive Ankle Work
Description: This is the amount of positive work performed by the ankle during walking normalized by body mass.
Time Frame: Same day; pre-stimulation (volitional) and post-stimulation (FES), day of the study
Population: Volitional and FES data available for participants with hemiparesis.
Measure: Mean (Standard Deviation); unit: Joules/body mass in kilograms
Arm/Group | Arm 1: FES
Number analyzed (Participants) | 8
Joules/body mass in kilograms
  Volitional | 0.1097 (0.0909)
  FES: Open loop | 0.1423 (0.1122)
  FES: Foot switch Trigger | 0.0869 (0.0447)

4. Secondary Outcome: The Impulse of the Anterior Ground Reaction Force Normalized by Body Mass.
Description: The is the magnitude of ground reaction force over time per step in the anterior direction during walking.
Time Frame: Same day: pre-stimulation (volitional) and post-stimulation (FES), day of the study
Population: Volitional and FES data available for participants with hemiparesis.
Measure: Mean (Standard Deviation); unit: Newtons*seconds/body mass in kilograms
Arm/Group | Arm 1: FES
Number analyzed (Participants) | 8
Newtons*seconds/body mass in kilograms
  Volitional | 0.0100 (0.0081)
  FES: Open loop | 0.0106 (0.0081)
  FES: Foot switch Trigger | 0.0109 (0.0102)

ADVERSE EVENTS:
Arm/Group | Arm 1: FES
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes